CLINICAL TRIAL: NCT01504607
Title: Corneal Endothelial Morphologic Assessment in Pediatric Cataract Surgery With IOL Implantation: Comparison of Preoperative and Early Postoperative Specular Microscopy
Brief Title: Corneal Endothelial Changes Following Pediatric Cataract Surgery With IOL Implantation
Status: Completed | Type: Observational
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: ICIRC-Pedspec; 2011-13 (Other: ICIRC)
Record Dates: First submitted 2011-12-27; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Congenital Cataract Surgery; IOL Implantation; Change in Corneal Endothelial Cell Morphology
Keywords: corneal endothelium; congenital cataract surgery; IOL implantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Congenital cataract surgery with IOL implantation: Congenital cataract surgery was performed with or without anterior vitrectomy, followed by in the bag IOL implantation
  Interventions: Procedure: Congenital Cataract Surgery

INTERVENTIONS:
Procedure: Congenital Cataract Surgery — Congenital cataract surgery with IOL implantation

SUMMARY:
Cataract surgery is known to cause loss of corneal endothelial cells. In adults, it is reported that anywhere between 2 to 15% loss of corneal endothelial cell density occurs following cataract surgery. However, no data is available regarding endothelial changes after cataract surgery with IOL implantation in pediatric eyes.

The aim of this study is to prospectively observe changes in endothelial cell density, coefficient of variation and hexagonality following cataract surgery with IOL implantation in pediatric eyes.

ELIGIBILITY:
Inclusion Criteria:

* Eyes undergoing pediatric cataract surgery with IOL implantation at Iladevi Cataract & IOL Research Center, Ahmedabad, India.
* Children older than 4 years undergoing cataract surgery with IOL implantation were included.

Exclusion Criteria:

* Exclusion criteria were as follows: eyes with traumatic or subluxated cataract and inability to get preoperative specular. Intraoperatively, sulcus fixated IOLs, and eyes with no IOL implantation were excluded.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children older than 4 years undergoing cataract surgery with IOL implantation were included.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial morphology | preoperatively to 3 months postoperatively
  Change in corneal endothelial cell density, (CD), coefficient of variation (CV) and % of hexagonality (6A) were studied from preoperatively to 3 months postoperatively

SECONDARY OUTCOMES:
Change in central corneal thickness | preoperatively to 3 months postoperatively
  Change in central corneal thickness from preop to 3 months postop was studied

REFERENCES:
- [Derived] Vasavada AR, Praveen MR, Vasavada VA, Shah SK, Vasavada V, Trivedi RH. Corneal endothelial morphologic assessment in pediatric cataract surgery with intraocular lens implantation: a comparison of preoperative and early postoperative specular microscopy. Am J Ophthalmol. 2012 Aug;154(2):259-265.e1. doi: 10.1016/j.ajo.2012.02.018. Epub 2012 Apr 27. PMID 22541660